CLINICAL TRIAL: NCT05610397
Title: Multicenter, Retrospective, Observational Clinical Study to Evaluate Clinical Outcome Measures and Safety Profiles for Patients With SDDD Treated With STALIF® C, or M, Ti or FLX Implants for 1 and 2 Levels.
Brief Title: Retrospective Study With Patients Treated With STALIF® C or M and Ti or FLX Implants for 1 and 2 Levels
Acronym: Stalif
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centinel Spine (Industry)
Responsible Party: Sponsor
Other Study IDs: VAL-P-0109
Record Dates: First submitted 2022-10-28; First posted 2022-11-09 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-11

CONDITIONS: Degenerative Disc Disease; Grade 1 Spondylolisthesis; Retrolisthesis; Symptomatic Cervical Disc Disease
Keywords: Retrolisthesis; Grade 1 Spondyloisthesis; Degenerative Disc Disease; Symptomatic Cervical Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (8):
- 1 level STALIF® C Ti: 25 patients who have a 1 level implant with STALIF® C Ti
  Interventions: Device: STALIF®
- 1 level STALIF® C FLX: 25 patients who have a 1 level implant with STALIF® C FLX
  Interventions: Device: STALIF®
- 1 level STALIF® M Ti: 25 patients who have a 1 level implant with STALIF® M Ti
  Interventions: Device: STALIF®
- 1 level STALIF® M FLX: 25 patients who have a 1 level implant with STALIF® M FLX
  Interventions: Device: STALIF®
- 2 level STALIF® C Ti: 25 patients who have a 2 level implant with STALIF® C Ti
  Interventions: Device: STALIF®
- 2 level STALIF® C FLX: 25 patients who have a 2 level implant with STALIF® C FLX
  Interventions: Device: STALIF®
- 2 level STALIF® M Ti: 25 patients who have a 2 level implant with STALIF® M Ti
  Interventions: Device: STALIF®
- 2 level STALIF® M FLX: 25 patients who have a 2 level implant with STALIF® M FLX
  Interventions: Device: STALIF®

INTERVENTIONS:
Device: STALIF® — STALIF® C, or M, Ti or FLX
  Other Names: STALIF® Cervical, Midline, Lumbar

SUMMARY:
This is a Retrospective, Observational Multi-Center study, utilizing patients diagnosed with up to a Grade1 spondylolisthesis or retrolisthesis or symptomatic degenerative disc disease and treated with STALIF® C, or M, Ti and/or FLX implants at one or two levels.

DETAILED DESCRIPTION:
The study is intended to codify the performance of the STALIF family of products. Its design is to provide retrospective data derived from the patient's medical and surgical chart and prospectively assess the treating surgeon and patient on their level of satisfaction post-operative up to present.

All subjects who sign an informed consent will be included in the prospective data collection via chart review at the individual investigational sites. The prospective data will come from subjects who complete the designated patient assessments as well as the treating surgeon. The data collection period will include surgeries performed between 2014 to present.

The analysis will support the safety profile of the product family and allow for comparison to the available literature as well as between device types (Ti versus FLX). Furthermore, data from this study will support post-market surveillance requirements for the STALIF family of products.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with up to a Grade1 spondylolisthesis or retrolisthesis or degenerative disc disease of the cervical or lumbar spine at time of surgery.
* 2 levels, between:

  * C: C2-T1 (neck)
  * M: L2-S1 (low back)
* Skeletally mature at the time of surgery with clinical and radiological evidence of degenerative disc disease of the cervical or lumbar spine.

Exclusion Criteria:

* Subject who had surgery with the STALIF devices at more than 2-levels.
* In the Investigator's opinion, the subject diagnosed with a disease or condition, which precludes the possibility of healing at the time of surgery

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgeon medical records. Hospital medical records.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-24 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) Questionnaire | Change from baseline at 24 months
  Assessing low back disability. Questionnaire consists of 10 sections with 6 possible choices in each section. Patient to choose 1 answer that best describes his/her ability to manage everyday activities. The questions weighted and summarized providing physical and mental health scores (PCS and MCS) ranging from 0 to 100. High scores indicating worse outcome and lower scores indicating better outcomes.
Neck Disability Index (NDI) | Change from baseline at 24 months
  Assessing cervical neck disability questionnaire. Questionnaire consists of 10 sections with 6 possible choices in each section. Patient to choose 1 answer that best describes his/her ability to manage everyday life activities. The questions weighted and summarized providing physical and mental health scores (PCS and MCS) and range from 0 to 100. High scores indicating worse outcome and lower scores indicating better outcomes.

SECONDARY OUTCOMES:
Patient Self Satisfaction Survey | Post-op at 24 months
  Self reported patient satisfaction survey consisting of 4 questions with 5 possible choices in each section. Patient to select one answer in each section. Scoring range from 0 to 100. Higher score extremely satisfied and lower score equals extremely dissatisfied.
Surgical Interventions | Post-op Day 1 of surgery to 6 months
  No secondary surgical interventions.
Adverse Events | Day of surgery to 12 months
  Adverse events
Surgeon Self Satisfaction Survey | Post-op at 24 months
  Surgeon Self Satisfaction Survey consists of 5 questions with 5 possible choices in each section. Surgeon to select one answer in each section. Scoring range from 0 to 100. Higher score extremely satisfied and lower score equals extremely dissatisfied.
Quality of Lift Questionnaire (SF-12) Prospective Arm of Study | Post-op at 24 months.
  SF-12 consists of 12 questions. Responses scored and summarized into physical and mental health composite scores (PCS and MCS) and range from 0 to 100. Higher score indicating better health. Score of 0 is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Illerhaus, MD, Principal Investigator — Orthopädisch-Neurochirurgisches Zentrum

IPD SHARING:
Plan to Share IPD: No
Retrospective Chart Review Study with a Prospective Arm. Surgery occurred between 2014 - present.